CLINICAL TRIAL: NCT01822223
Title: A Controlled, Double-Blind, Randomized, Parallel-Arm, Clinical Trial to Evaluate the Effectiveness of Laser-Ablated Implant-Abutments for Enhanced Oral Mucosal Healing
Brief Title: A Study to Evaluate the Effectiveness of Laser-Ablated Implant-Abutments to Promote Tissue Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: BioHorizons, Inc. (Industry)
Responsible Party: Principal Investigator, Michael Reddy, DMD, Professor, Dean, School of Dentistry, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Bio-LL-001
Record Dates: First submitted 2013-02-27; First posted 2013-04-02 (Estimated); Results first posted 2017-01-25 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2016-09

CONDITIONS: Jaw, Edentulous, Partially
Keywords: Dental Implants; Implant abutments
MeSH Terms: conditions — Jaw, Edentulous, Partially

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laser-ablated dental implant-abutments (Experimental): Laser-ablated dental implant abutments will be attached to surgically placed dental implants.
  Interventions: Device: Dental implant-abutments
- Smooth implant-abutments (Active Comparator): Smooth dental implant-abutments will be attached to surgically placed dental implants.
  Interventions: Device: Dental implant-abutments

INTERVENTIONS:
Device: Dental implant-abutments — At week-8, abutments will be removed and replaced with new Laser-Lok® abutments. An inter-arm randomization will assign subjects to one of two sub-groups per treatment arm. Sub-groups 1-a & 2-a: will receive a new Laser-Lok® abutment and a soft-tissue biopsy at week-8; a force-probe clinical attachment assessment of the same site will be delayed until week-16.
  Sub-groups 1-b & 2-b: will receive a new Laser-Lok® abutment and a force-probe clinical attachment assessment at week-8; a biopsy harvested from the same study site will be delayed until week-16.
  The implants will be restored following standard technique and a final visit will occur 6 months following permanent restoration.
  Other Names: BioHorizons' Laser-Lok® abutment; BioHorizons' smooth-surfaced abutment

SUMMARY:
The purpose of this study is to determine which implant-abutment design is more likely to promote early soft-tissue healing processes and/or will enhance longitudinal peri-implant bone and soft-tissue health.

DETAILED DESCRIPTION:
The study will assess the integrity of the peri-implant oral soft-tissue attachment to implant abutments by comparing tissue responses to a laser-ablated implant-abutment and an implant-abutment manufactured with a smooth surface.

Investigators will assess the initial post-surgical peri-implant attachment-seal and will test whether or not the tissue-abutment interface re-forms with equal integrity when the abutment is removed and replaced with a new abutment.

Data will include histological, radiographic, clinical, and subjective aesthetics to compare the effectiveness of two abutment designs. Both devices are supplied by the BioHorizons Implant Systems Inc. of Birmingham, Alabama; the abutments are analogous in design and material except the test device has a laser-ablated surface and the control abutment is smooth.

ELIGIBILITY:
Inclusion Criteria:

1. At least 19 years old
2. Healthy enough to under go treatment
3. Have one or more edentulous sites that exhibit adequate natural bone and sufficient keratinized tissue
4. Demonstrated willingness to undergo study treatment and to comply with study timeline -

Exclusion Criteria:

1. Full edentulism
2. Any chronic health condition or medication that in the opinion of the investigators may adversely affect bone healing
3. Any indication of an inability to make autonomous decisions

   -

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-11; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Reddy, DMD, DMSc, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham School of Dentistry, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Geurs NC, Geisinger ML, Vassilopoulos PJ, O'Neal SJ, Haigh SJ, Reddy MS. Optimizing Connective Tissue Integration on Laser-Ablated Implant Abutments. Clin Adv Periodontics. 2016 Aug;6(3):153-159. doi: 10.1902/cap.2016.150068. PMID 31535464

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Laser-ablated Dental Implant-abutments | Smooth Implant-abutments
Started | 10 | 10
Completed | 10 | 9
Not Completed | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Laser-ablated Dental Implant-abutments: Laser-ablated dental implant abutments will be attached to surgically placed dental implants.
  Dental implant-abutments: At week-8, abutments will be removed and replaced with new Laser-Lok® abutments. An inter-arm randomization will assign subjects to one of two sub-groups per treatment arm. Sub-groups 1-a & 2-a: will receive a new Laser-Lok® abutment and a soft-tissue biopsy at week-8; a force-probe clinical attachment assessment of the same site will be delayed until week-16.
  Sub-groups 1-b & 2-b: will receive a new Laser-Lok® abutment and a force-probe clinical attachment assessment at week-8; a biopsy harvested from the same study site will be delayed until week-16.
  The implants will be restored following standard technique and a final visit will occur 6 months following permanent restoration.
- Smooth Implant-abutments: Smooth dental implant-abutments will be attached to surgically placed dental implants.
  Dental implant-abutments: At week-8, abutments will be removed and replaced with new Laser-Lok® abutments. An inter-arm randomization will assign subjects to one of two sub-groups per treatment arm. Sub-groups 1-a & 2-a: will receive a new Laser-Lok® abutment and a soft-tissue biopsy at week-8; a force-probe clinical attachment assessment of the same site will be delayed until week-16.
  Sub-groups 1-b & 2-b: will receive a new Laser-Lok® abutment and a force-probe clinical attachment assessment at week-8; a biopsy harvested from the same study site will be delayed until week-16.
  The implants will be restored following standard technique and a final visit will occur 6 months following permanent restoration.
- Total: Total of all reporting groups
Arm/Group | Laser-ablated Dental Implant-abutments | Smooth Implant-abutments | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Gender [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number od Participants With Consistent Connective Tissue Integration at a Histologic Level
Description: Connective tissue integration was assessed by radio graphic images of tissue and bone surrounding the implant.
Time Frame: 8 weeks post-abutment placement
Population: The number of participants entered represents measured data.
Measure: Number; unit: participants
Arm/Group | Laser-ablated Dental Implant-abutments | Smooth Implant-abutments
Number analyzed (Participants) | 10 | 10
participants | 10 | 10

2. Secondary Outcome: Grams of Force Needed to Disrupt Tissue Attachment to the Abutment
Description: A force transducing periodontal probe instrument will electronically capture the grams of force needed to disrupt the attachment to the implant abutment; tissues will be probed from the gingival margin to the alveolar bone crest at 4 points around each abutment and an adjacent tooth: measurements will be captured from the mesial, buccal, distal, and lingual. The specific force probe generates a descriptive graph that demonstrates the cumulative force and distribution necessary to disrupt the attachment of the gingival tissues to the abutment. These graphs were recorded, but were difficult to interpret and have not been reported.
Time Frame: 8 weeks post-abutment placement
Population: No data was collected on subjects from the mesial, buccal, distal or lingual sites as sites were not assessed on subjects for reasons unknown.
Arm/Group | Laser-ablated Dental Implant-abutments | Smooth Implant-abutments
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Mean Change in Millimeters of Clinical Attachment to the Abutment
Description: A periodontal probe will be used to measure the level of clinical attachment to the abutment in millimeters. Measurements will be captured at 4 points around each abutment; mesial, buccal, distal, and lingual. All measurements were considered and the change in attachment level was assessed at each individual site. Data were reported as descriptive and were used to elucidate potential advantages and/or disadvantages of varying abutment types. These data were strictly confirmatory to the proof-in-principle histology presented in the report. Measures were taken at 8 weeks, 12 weeks, 16 weeks and 12 months to determine if attachment to one abutment type was more or less stable over time. The specific force probe generates a descriptive graph that demonstrates the cumulative force and distribution necessary to disrupt the attachment of the gingival tissues to the abutment. These graphs were recorded, but were difficult to interpret and have not been reported.
Time Frame: 8 weeks post-abutment placement
Population: as for outcome 2
Arm/Group | Laser-ablated Dental Implant-abutments | Smooth Implant-abutments
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Mean Change in Millimeters of Clinical Attachment to the Abutment
Description: as for outcome 3
Time Frame: 12 weeks post-abutment placement
Population: as for outcome 2
Arm/Group | Laser-ablated Dental Implant-abutments | Smooth Implant-abutments
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Mean Change in Millimeters of Clinical Attachment to the Abutment
Description: as for outcome 3
Time Frame: 16 weeks post-abutment placement
Population: as for outcome 2
Arm/Group | Laser-ablated Dental Implant-abutments | Smooth Implant-abutments
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Mean Change in Millimeters of Clinical Attachment to the Abutment
Description: as for outcome 3
Time Frame: 12 month post-abutment placement
Population: as for outcome 2
Arm/Group | Laser-ablated Dental Implant-abutments | Smooth Implant-abutments
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from time of enrollment, January 5, 2011 to close of study, September 12, 2014.
Arm/Group | Laser-ablated Dental Implant-abutments | Smooth Implant-abutments
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes